CLINICAL TRIAL: NCT07056335
Title: Physical Activity and Percussive Massage Therapy for Reducing Pain in Older Women
Acronym: MAPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Shiyu Li, Postdoctoral Research Fellow, Motivation Lab School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: HUM00262006
Record Dates: First submitted 2025-06-13; First posted 2025-07-09 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Pain, Chronic
Keywords: behavior change
MeSH Terms: conditions — Chronic Pain | interventions — Blood Glucose Self-Monitoring; Exercise

STUDY DESIGN:
Intervention Model Description: This is a 2 (self-monitoring PA: daily prompts vs none) x 2 (self-monitoring PMT: daily prompts vs none) factorial experiment with random assignment. All participants will receive a Theragun® device and education about the benefits of PA and PMT for older adults. Participants will then be randomly assigned to one of four experimental groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessor will not know which group the participants are assigned to. Instead, the assigned group is be as numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical Activity Self-monitoring (Experimental): Participants will receive a Theragun® device and education about the benefits of PA and PMT for older adults.
  Participants will receive daily email for physical activity self-monitoring.
  Interventions: Behavioral: Self-monitoring; Behavioral: Physical activity and percussive massage therapy education; Device: Percussive massage therapy
- Percussive Massage Therapy Self-monitoring (Experimental): Participants will receive a Theragun® device and education about the benefits of PA and PMT for older adults.
  Participants will receive daily email for massage gun usage self-monitoring.
  Interventions: Behavioral: Self-monitoring; Behavioral: Physical activity and percussive massage therapy education; Device: Percussive massage therapy
- Physical activity and Percussive Massage Therapy Self-monitoring (Experimental): Participants will receive a Theragun® device and education about the benefits of PA and PMT for older adults.
  Participants will receive daily email for physical activity and massage gun usage self-monitoring.
  Interventions: Behavioral: Self-monitoring; Behavioral: Physical activity and percussive massage therapy education; Device: Percussive massage therapy
- No self-monitoring (Active Comparator): Participants will receive a Theragun® device and education about the benefits of PA and PMT for older adults.
  Interventions: Behavioral: Physical activity and percussive massage therapy education; Device: Percussive massage therapy

INTERVENTIONS:
Behavioral: Self-monitoring — Self-monitoring as a behavior change technique to support pain self-care behaviors
  Arms: Percussive Massage Therapy Self-monitoring; Physical Activity Self-monitoring; Physical activity and Percussive Massage Therapy Self-monitoring
Behavioral: Physical activity and percussive massage therapy education — Participants will receive education on why physical activity and massage are important for pain self-care. They will also receive daily physical activity and massage goals.
Device: Percussive massage therapy — Participants will receive a massage gun to support daily pain self-care.
  Other Names: Massage gun

SUMMARY:
Over 60% of women aged 65 and older suffer from pain, yet this group is underrepresented in research. Physical activity and percussive massage therapy may help manage pain, but both require consistent engagement, making long-term participation challenging for most people. Self-monitoring could improve adherence to these pain management efforts, but the optimal strategies for self-monitoring remain unknown.

This is a a 2x2 factorial randomized controlled trial in older women (N = 108) to determine which behavior(s) should be self-monitored to (1) promote engagement in physical activity and percussive massage therapy and (2) reduce pain. This study design will allow examination on effects of self-monitoring across different behaviors to identify the most effective strategies for improving pain management adherence and reducing pain.

DETAILED DESCRIPTION:
Pain is a common and disabling condition, affecting 1.5 billion people worldwide. Chronic pain is especially prevalent in women and older adults; over 63% of women aged 65+ report chronic pain. Yet this population has been understudied. Two evidence-based strategies hold promise for managing pain in older women: physical activity (PA) and percussive massage therapy (PMT).

PA is widely recommended for pain relief and improving functioning in older adults. However, pain is a commonly-cited barrier to PA. PMT through a massage gun offers promise for both acute pain management and reducing pain as a barrier to physical activity. PMT may be useful, however, few studies have examined the effectiveness of PMT for pain relief in older women, either alone or in combination with physical activity. PA and PMT also share a common challenges as pain management strategies - both require consistent engagement, yet long-term participation is challenging for most people.

Self-monitoring, the practice of recalling and recording a desired behavior regularly, is a widely adopted, evidence-based technique that supports behavior change. Conceptually, self-monitoring of PA and PMT should increase engagement in those behaviors and reduce pain. Yet, self-monitoring can be burdensome and difficult to maintain. Previous research found that engagement in self-monitoring within the first month may have long-lasting effects, but individuals typically disengage during early weeks. Therefore, limiting the scope of self-monitoring burden is important for long-term adherence. This research will answer the question, "Should a daily self-monitoring intervention focus on PA, PMT or both to promote engagement in those behaviors and reduce pain intensity and interference in older women?" There are two specific aims of this study:

Aim 1 (Behavior Change). To determine which behavior(s) should be self-monitored in an intervention to promote engagement in PA and PMT.

Aim 2 (Pain). To determine which behavior(s) should be self-monitored in an intervention to reduce pain intensity and interference.

ELIGIBILITY:
Inclusion Criteria:

1. Older aged female (65 years of age or older)
2. Self-report pain as a barrier to PA
3. Self-report not engaging in regular aerobic physical activity
4. Express an interest in increasing PA levels.
5. Proficient in English
6. Own an IOS or Android smartphone with regular internet access
7. Check emails at least daily
8. Capable of providing informed consent
9. Willing to use a massage gun for 3 months
10. Live in continental US

Exclusion Criteria:

1. Planned surgery that limits mobility in the next 2 months.
2. Concurrently participating in other pain management or physical activity programs
3. Cancer-related pain
4. Neurological disorder that affects cognition
5. Mobility impairments that prevent unassisted walking.
6. Receiving active medical treatment that would impair protocol compliance

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Self-reported pain intensity and interference | Baseline, 1 month, 2 month
  Self-reported pain will be assessed using Brief Pain Inventory. The Brief Pain Inventory is a self-report measure that assesses both pain severity and the degree to which pain interferes with daily functioning. Scores are reported on a numeric rating scale ranging from 0 to 10, with higher scores indicating worse outcomes. Specifically, 0 represents "no pain" or "no interference," while 10 represents "pain as bad as you can imagine" or "complete interference." The Brief Pain Inventory yields two main scores: a Pain Severity score, calculated as the mean of four items assessing worst, least, average, and current pain; and a Pain Interference score, calculated as the mean of seven items assessing interference with general activity, mood, walking ability, work, relationships, sleep, and enjoyment of life.

SECONDARY OUTCOMES:
Average Daily Step Counts | Baseline, 1 month, 2 month
  Average daily step counts recorded by Actigraph accelerometer over a 7-day monitoring period

OTHER OUTCOMES:
Self-monitoring engagement | Daily over the first month
  Self-monitoring engagement will be assessed as a daily binary outcome (yes/no) over the first month of the study. Participants will receive daily email surveys prompting them to log the duration of time spent in each physical activity intensity level and/or the duration of self-massage for five targeted muscle groups (calves, glutes, hamstrings, quadriceps, and lower back). The unit of measure will be the percentage of days on which participants completed the self-monitoring prompt, as indicated by a "yes" response to the daily survey.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyu Li, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No